CLINICAL TRIAL: NCT05235932
Title: A Prospective, Multicenter, Randomized, Controlled Study of the Clinical Efficacy of Robotic and Laparoscopic Radical Total Gastrectomy in Locally Advanced Middle and Upper Gastric Cancer
Brief Title: the Clinical Efficacy of Robotic and Laparoscopic Radical Total Gastrectomy in Locally Advanced Middle and Upper Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Collaborators: Chinese PLA General Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Lanzhou Military Region General Hospital (Unknown); Gansu Provincial Hospital (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Guangxi Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Xiangya Hospital of Central South University (Other); Hebei Medical University Fourth Hospital (Other); The Affiliated Hospital of Qingdao University (Other); The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02
Record Dates: First submitted 2022-02-10; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer; Robotic Gastrectomy
Keywords: robotic radical total gastrectomy; Gastric Cancer; laparoscopic radical total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic radical total gastrectomy with D2 lymphadenectomy (Experimental): After exploration and randomization, patients received robotic radical total gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Robotic radical total gastrectomy with D2 lymphadenectomy
- Laparoscopic radical total gastrectomy with D2 lymphadenectomy (Active Comparator): After exploration and randomization, patients received laparoscopic radical total gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Laparoscopic radical total gastrectomy with D2 lymphadenectomy

INTERVENTIONS:
Procedure: Robotic radical total gastrectomy with D2 lymphadenectomy — Most surgical procedures are performed using the robot system.
  Arms: Robotic radical total gastrectomy with D2 lymphadenectomy
Procedure: Laparoscopic radical total gastrectomy with D2 lymphadenectomy — Without the robot system, Most surgical procedures are performed using laparoscopic equipment.
  Arms: Laparoscopic radical total gastrectomy with D2 lymphadenectomy

SUMMARY:
To evaluate the clinical efficacy (safety, feasibility and long-term efficacy) of robotic radical total gastrectomy and laparoscopic radical total gastrectomy in patients with locally advanced middle and upper gastric adenocarcinoma (CT2-4A, N-/+, M0) .

DETAILED DESCRIPTION:
In the field of gastrectomy, Hashizume et al. first reported robotic gastrectomy in 2002. Since then, reports on the safety and feasibility of the application of robotic surgical system in the treatment of gastric cancer (GC) have gradually increased. Reports of robotic surgery for GC are increasing, especially in Asia. Several studies confirmed the advantages of robotic gastrectomy when compared with laparoscopic gastrectomy. However, whether robotic radical total gastrectomy is noninferior to laparoscopic radical total gastrectomy remains unclear. The investigator first carried out this study in the world to evaluate the efficacy of robotic radical total gastrectomy versus laparoscopic radical total gastrectomy for GC.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age between 18 and 75 years 2.The primary gastric lesion was histopathologically diagnosed as middle and upper gastric adenocarcinoma (papillary adenocarcinoma PAP, tubular adenocarcinoma TUB, mucinous adenocarcinoma MUC, signed-ring cell carcinoma SIG, poorly differentiated adenocarcinoma POR) by endoscopic biopsy.

  3.Preoperative clinical stages were CT2-4A、 N-/+、and M0 (according to AJCC-8th TNM tumor staging) 4.Excepting to perform radical total gastrectomy and D2 lymph node dissection can achieve R0 resection.

  5.American Society of Anesthesiology (ASA) score class I, II, or III 6.Written informed consent

Exclusion Criteria:

1. Preoperative examination suggested disease staging cT1, N-/+, and M0 (according to AJCC-8th TNM tumor staging )
2. Women during pregnancy or breast-feeding
3. Severe mental disorder
4. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
5. History of previous gastrectomy(except for ESD/EMR for gastric cancer )
6. Enlarged or bulky regional lymph node over 3 cm by preoperative imaging
7. History of other malignant disease within the past five years
8. History of previous neoadjuvant chemotherapy or radiotherapy
9. History of unstable angina or myocardial infarction within past six months
10. History of cerebrovascular accident within past six months
11. History of continuous systematic administration of corticosteroids within one month
12. Requirement for simultaneous surgery for other disease(except laparoscopic cholecystectomy)
13. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
14. FEV1 (forced expiratory volume in one second)<50% of predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  3-year disease free survival rate

SECONDARY OUTCOMES:
Morbidity rates | 30 days
  This is for the early postoperative complication, which defined as the event observed within 30 days after surgery.
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
overall postoperative serious morbidity rates | 30 days
  Refers to the incidence of early postoperative complication which is graded as Clavien-Dindo IIIA or higher
Total Number of Retrieved Lymph Nodes | 1 day
  Total Number of Retrieved Lymph Nodes
postoperative recovery course | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
postoperative nutritional status | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
inflammatory immune response | Preoperative 3 days and postoperative 1, 3, and 5 days
  The variation of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response

CONTACTS AND LOCATIONS:
Overall Officials: Chang-ming Huang, MD, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China